CLINICAL TRIAL: NCT05374096
Title: The Effect of Music on Pain in Patients Undergoing Ventral Hernia Repair With Mesh: A Double-Blind Randomized Controlled Trial
Brief Title: Study Exploring the Effect of Music on Pain After Ventral Hernia Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Ajita Prabhu, MD, Staff Physician, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-286
Record Dates: First submitted 2022-05-02; First posted 2022-05-16 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Postoperative Pain, Acute; Ventral Hernia; Hernia Abdominal Wall; Surgery; Anxiety
Keywords: Music
MeSH Terms: conditions — Pain, Postoperative; Hernia, Ventral; Hernia, Abdominal; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Via Headphones (Experimental): Headphones will be placed with patient-selected music playing for the duration of the surgical procedure.
  Interventions: Other: Patient-Chosen Music
- Silence Via Headphones (Control) (Placebo Comparator): Headphones will be placed with silence for the duration of the surgical procedure.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Patient-Chosen Music — Music played into headphones.
  Arms: Music Via Headphones
Other: Placebo — Silence into headphones.
  Arms: Silence Via Headphones (Control)

SUMMARY:
The purpose of this study is to assess whether listening to music during surgery has an effect on pain or anxiety after surgery.

DETAILED DESCRIPTION:
After being informed about the study and potential risks and meeting eligibility criteria, all patients giving written informed consent will be scheduled for their hernia repair surgery. On the day of surgery, patients will be randomized in a double-blind manner (participant and investigator) in a 1:1 ratio to listen to patient-chosen music during their surgery via headphones or just listen to silence via headphones. Pain and anxiety will then be assessed after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Adults having open retromuscular ventral hernia repair with mesh, with or without myofascial release for a hernia width ≤ 20 cm
2. Adults having open flank hernia repair that requires a myofascial release with mesh
3. Adults having parastomal hernia repair with mesh

Exclusion Criteria:

1. Primary language other than English, or lack of English language fluency
2. Hearing impairment, with or without use of hearing aids
3. Neurologic condition that, in the opinion of the investigators, may preclude accurate assessment of postoperative pain and anxiety
4. Patients who will remain intubated after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 321 (Actual)
Dates: Start 2022-06-13 (Actual); Primary Completion 2023-07-15 (Actual); Study Completion 2023-07-17 (Actual)

PRIMARY OUTCOMES:
Post operative Pain | At 24 hours (+- 3 hours) after surgery end time.
  Pain scores will be assessed using the Numeric Pain Rating Scale (NRS-11); The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")

SECONDARY OUTCOMES:
Post operative Anxiety | At 24 hours (+- 3 hours) after surgery end time.
  Anxiety scores will be assessed using State Trait Anxiety Index-6 (STAI-6) Anxiety tool (a 6 question patient-reported anxiety assessment). The higher the total, the greater the anxiety is.

OTHER OUTCOMES:
Post operative Pain - 3 days | Collected at 3 time points after surgery end time - 24 hours (+- 3 hours), 48 hours (+-3 hours) and 72 hours (+-3 hours)
  Pain scores will be assessed using the Numeric Pain Rating Scale (NRS-11); The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
Post operative Pain - cumulative | Will be collected repeatedly by nursing staff per nursing protocol for the first 24 hours after surgery end time.
  Pain scores will be assessed using the Numeric Pain Rating Scale (NRS-11); The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable")
Post operative Anxiety - 3 days | Collected at 3 time points after surgery end time - 24 hours (+- 3 hours), 48 hours (+-3 hours) and 72 hours (+-3 hours)
  Anxiety scores will be assessed using State Trait Anxiety Index-6 (STAI-6) Anxiety tool (a 6 question patient-reported anxiety assessment). The higher the total, the greater the anxiety is.
Post operative opioid consumption | During the first 72 hours after surgery end time.
  Cumulative opioid consumption converted into morphine milligram equivalents.
Intraoperative sedative use | From induction of anesthesia to arrival in the post anesthesia care unit on the day of procedure
  Total number of intravenous and inhaled anesthetics, benzodiazepines, and opioid medications.

CONTACTS AND LOCATIONS:
Overall Officials: Ajita Prabhu, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Main Campus, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Maskal SM, Gentle CK, Ellis RC, Tu C, Rosen MJ, Petro CC, Miller BT, Beffa LRA, Chang JH, Messer N, Melland-Smith M, Jeekel J, Prabhu AS. Does selective intraoperative music reduce pain following abdominal wall reconstruction? A double-blind randomized controlled trial. Hernia. 2024 Oct;28(5):1831-1841. doi: 10.1007/s10029-024-03092-y. Epub 2024 Jun 18. PMID 38890182